CLINICAL TRIAL: NCT05068882
Title: Impact of Preoperative Oral Diets on Postoperative Fluid Collection After Axillary Lymphadenectomy
Brief Title: Impact of Oral Diets on Postoperative Fluid Collection
Acronym: BC1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stanley Dudrick's Memorial Hospital (Other)
Responsible Party: Principal Investigator, Stanislaw Klek, Head of the Unit, Stanley Dudrick's Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC1
Record Dates: First submitted 2021-09-25; First posted 2021-10-06 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Immunonutrition Diet

STUDY DESIGN:
Intervention Model Description: 4 arm randomized study
Who Masked: Investigator, Outcomes Assessor
Masking Description: The physician is unaware of the type of the intervention. The type of intervention is given by the independent person to dietitian instructing the patient how to use the product.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Immunonutrition (Experimental): Oral immunonutrition containing arginine, omega-PUFAs and antioxidants
  Interventions: Dietary Supplement: Immunonutrition
- High-protein diet (Active Comparator): Oral nutrition with high-protein content
  Interventions: Dietary Supplement: High-protein nutrition
- Standard nutrition (Active Comparator): Oral nutrition with standard ingredients
  Interventions: Dietary Supplement: Standard nutrition
- No intervention (No Intervention): No intervention

INTERVENTIONS:
Dietary Supplement: Immunonutrition — Oral immunonutrition containing arginine, omega-PUFAs and antioxidants
  Arms: Immunonutrition
Dietary Supplement: High-protein nutrition — Oral nutrition with high-protein content
  Arms: High-protein diet
Dietary Supplement: Standard nutrition — Oral nutrition with standard ingredients
  Arms: Standard nutrition

SUMMARY:
Patients after the surgical removal of axillary lymphnodes suffers from prolonged fluid collections. The aim of the study is to assess the impact of oral immunonutrition and high-protein diets on the reduction of fluid collection.

DETAILED DESCRIPTION:
Patients after the surgical removal of axillary lymphnodes suffers from prolonged fluid collections, which requires either prolonged drainage or multiple punctuations. The aim of the study is to assess the impact of oral immunonutrition and high-protein diets on the reduction of fluid collection.

ELIGIBILITY:
Inclusion Criteria:

* confirmed breast cancer or melanoma
* scheduled surgery with axillary lymph nodes resection
* informed consent
* eligible for surgery

Exclusion Criteria:

* benign disease
* no consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Fluid collection | 6 months
  The volume of fluid collection after lymph nodes resection expressed in mililiters

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw Klek, PhD, Principal Investigator — Stanley Dudrick's Memorial Hospital
Locations (2):
- Poland (2):
  - Maria Sklodowska-Curie National Cancer Institute, Krakow, Malopolska
  - Stanley Dudrick's Memorial Hospital, Skawina

IPD SHARING:
Plan to Share IPD: No